CLINICAL TRIAL: NCT01884571
Title: A Novel Immunosuppression Intervention for the Treatment of Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Immunosuppression in Amyotrophic Lateral Sclerosis (ALS)
Acronym: NIPALS2013
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Jonathan D. Glass, M.D., Director, Emory ALS Clinic, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00064218; NIP-ALS-2013 (Other: Other); 2013P000981 (Other: Other)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Immunosuppression; ALS; Neuromuscular Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases | interventions — Basiliximab; Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisone; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immunosuppression Regimen (Experimental): Basiliximab Methylprednisolone Prednisone Tacrolimus Mycophenolate mofetil
  Interventions: Drug: Basiliximab; Drug: Methylprednisolone; Drug: Prednisone; Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Basiliximab — 20 mg, IV (in the vein) on day 1 and 4.
  Other Names: Simulect
Drug: Methylprednisolone — 125 mg, IV (in the vein) on day 1.
  Other Names: Solumedrol
Drug: Prednisone — 60 mg PO (by mouth) on days 2-7, 40 mg PO days 8-14, 20 mg PO days 15-21, and 10mg PO days 22-28.
  Other Names: Deltasone; Orasone
Drug: Tacrolimus — 1-5 mg PO, twice a day (BID) days 2-180.
  Other Names: Prograf
Drug: Mycophenolate mofetil — 500 mg PO, BID days 2-7, 500 mg PO each morning and 1000 mg each night, days 8-14, 1000 mg PO BID days 15-180.
  Other Names: Cellcept

SUMMARY:
This is a multicenter, 15-month study evaluating the effect of immunosuppression treatment on the rate of change on the ALS Functional Rating Scale (Revised) (ALSFRS-R) score in up to 33 subjects with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
In an ongoing safety trial of neural stem cell injections into the spinal cord of patients with ALS at Emory University, Atlanta, Georgia, one patient has demonstrated clear improvement by objective clinical and electrophysiological measures, a finding that is unheard of in patients with ALS.

This patient had an improvement in ALSFRS-R by 1.4 points per month. In 826 historical controls from the Northeast ALS Consortium (NEALS) and the Western ALS Consortium (WALS) database where ALSFRS-R was documented at 2 or more visits, there have been no patients that have shown improvement in ALSFRS as seen in this case. Additionally, 5 patients in the stem cell trial who were not on mechanical ventilators at the time of surgery seem to have very slow disease progression as compared to the expectation from current understanding of typical disease course. This observation raises consideration for a disease-modifying effect of the novel immunosuppression regimen used in this trial. Also, given that ALS is clinically an extraordinarily heterogeneous disease, the diagnosis of ALS may represent a group of phenotypically similar but pathogenically variable disorders. It is possible that there exists a subset of patients with an immune-responsive ALS subtype that has not been previously recognized.

Recent studies have furthered the understanding of the immune mechanisms that contribute to ALS progression. Microglia and lymphocytes have both neurotoxic and neuroprotective functions depending on activation states and physiologic conditions within the nervous system. Therefore, targeted immunotherapies that proportionally suppress neurotoxic immune elements, while sparing or promoting protective elements, seemingly have more potential to modify disease course in ALS than previously tested regimens. It is postulated that the immunosuppression treatment given to the stem cell patients may have exhibited neuroprotective effects by favorably promoting the ratio of regulatory T cells and other protective immune mediators in relation to neurotoxic immune modulators. It is hoped that this trial will optimize the chance of replicating these findings and advance knowledge about the complex changes that occur within the immune system in patients with ALS before and after treatment with an immunosuppression regimen.

The primary outcome measure will be rate of change of ALSFRS-R. A clinical response will be defined as a rate of change of ALSFRS-R of +6 points over a 6 month period (mean of change of +1 point per month).

Secondary outcome measures will include slow vital capacity (SVC), grip strength, and hand held dynamometry (HHD). The change in rate of progression in clinical measures will be monitored to look for a potential disease-modifying effect of the immunosuppression regimen. Blood and cerebrospinal fluid immune system markers will be also be studied.

If a clinical response is seen among study participants following treatment, further analyses will be conducted to explore any differential effects of immunosuppression in participants with early-stage disease and later-stage disease. To ensure adequate numbers of participants for conditional analyses stratifying by symptom onset date, participants will be enrolled based on symptom onset within 24 months of the screening visit or more than 24 months before screening. All participants will have the same treatment and will be treated as a single group for the analyses of the main study outcomes.

ELIGIBILITY:
Inclusion Criteria for participants with symptom onset within the past 24 months:

* Male or female patients 18-65 years of age.
* ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial Criteria.
* Symptom onset ≤ 24 months from screening visit.
* A score of ≥38 on the Revised ALS Functional Rating Scale.
* Slow vital capacity (SVC) measure >80% of predicted for gender, height and age at screening.
* Subjects must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days, prior to the screening visit (riluzole-naïve subjects are permitted in the study).
* Negative tuberculosis (TB) test within 3 months of Screening Visit.
* Subjects medically able to undergo lumbar puncture (LP) as determined by the investigator (i.e., no bleeding disorder, allergy to local anesthetics, or a skin infection at or near the LP site).
* Capable of providing informed consent and following study procedures.
* Women must not be able to become pregnant (e.g. post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study.
* Women of childbearing potential must have a negative pregnancy test at screening and be non-lactating.
* Geographic accessibility to the study site.

Inclusion Criteria for participants with symptom onset greater than 24 months before screening:

* Male or female patients age 18 or older.
* ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial Criteria.
* Symptom onset >24 months from screening visit.
* Subjects must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days, prior to the screening visit (riluzole-naïve subjects are permitted in the study).
* Negative tuberculosis (TB) test within 3 months of Screening Visit.
* Subjects medically able to undergo lumbar puncture (LP) as determined by the investigator (i.e., no bleeding disorder, allergy to local anesthetics, or a skin infection at or near the LP site).
* Capable of providing informed consent and following study procedures.
* Geographic accessibility to the study site.
* Women must not be able to become pregnant (e.g. post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study.
* Women of childbearing potential must have a negative pregnancy test at screening and be non-lactating.

Exclusion Criteria

* Prior use of basiliximab, solumedrol, prednisone, tacrolimus or mycophenolate mofetil within 30 days of the Screening Visit.
* Known allergy or sensitivity to basiliximab, solumedrol, prednisone, tacrolimus or mycophenolate mofetil or a formulation of one of these drugs.
* Treatment with an immunosuppressant medication within 30 days of the Screening Visit.
* Active peptic ulcer disease.
* Any medical disorder that would make immunosuppression contraindicated including, but not limited to, human immunodeficiency virus (HIV), tuberculosis, or evidence of active cytomegalovirus (CMV) or infection.
* Subjects who have a diaphragm pacing system (DPS).
* Women who are pregnant, breastfeeding, or planning to become pregnant in the next 12 months.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Use of invasive or non-invasive mechanical ventilation (including Continuous Positive Airway Pressure (CPAP) or Bi-level Positive Airway Pressure (BiPAP)) for any part of the day or night prior to the Screening Visit (participants with symptom onset within past 24 months only).
* Exposure to any other agent currently under investigation for the treatment of patients with ALS (off-label use or investigational) within 30 days of the Screening Visit.
* Inability to safely complete study activities based on the discretion of the site investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Glass, MD, Principal Investigator — Emory University; Christina N Fournier, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fournier CN, Schoenfeld D, Berry JD, Cudkowicz ME, Chan J, Quinn C, Brown RH, Salameh JS, Tansey MG, Beers DR, Appel SH, Glass JD. An open label study of a novel immunosuppression intervention for the treatment of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2018 May;19(3-4):242-249. doi: 10.1080/21678421.2017.1421666. Epub 2018 Jan 8. PMID 29308669
- See also: Northeast ALS Consortium Website — http://www.alsconsortium.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited for this study from three Northeast ALS Consortium (NEALS) centers in the USA (Emory University in Atlanta, Georgia, Massachusetts General Hospital in Boston, Massachusetts, and University of Massachusetts Medical School in Worcester, Massachusetts. Recruitment occurred between October 2013 and October 2014.
Groups:
- Immunosuppression Regimen: All participants received the same treatment intervention consisting of basiliximab, methylprednisolone, prednisone, tacrolimus and mycophenolate mofetil. Doses of each medication varied by the day of treatment (described below) and the treatment period lasted for six months.
  Basiliximab: 20 mg, IV (in the vein) on day 1 and 4.
  Methylprednisolone: 125 mg, IV (in the vein) on day 1.
  Prednisone: 60 mg PO (by mouth) on days 2-7, 40 mg PO days 8-14, 20 mg PO days 15-21, and 10mg PO days 22-28.
  Tacrolimus: 1-5 mg PO, twice a day (BID) days 2-180.
  Mycophenolate mofetil: 500 mg PO, BID days 2-7, 500 mg PO each morning and 1000 mg each night, days 8-14, 1000 mg PO BID days 15-180.
Period: Overall Study
Arm/Group | Immunosuppression Regimen
Started | 31
Completed | 23
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Groups:
- Immunosuppression Regimen: All participants received the same treatment intervention consisting of basiliximab, methylprednisolone, prednisone, tacrolimus and mycophenolate mofetil. Doses of each medication varied by the day of treatment and the treatment period lasted for six months.
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
Timing of Symptom Onset [Count of Participants; unit: Participants]
  Less than or equal to 24 months prior to screening | 20
  More than 24 months prior to screening | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Average Increase in ALSFRS-R Score of One Point Per Month
Description: The ALS Functional Rating Scale - Revised (ALSFRS-R) is an ordinal rating scale (0 through 4) used to determine the ALS patient's self assessment of their ability and need for assistance in 12 activities or functions. This is a validated scale, both in person and by phone, which provides a total score (best of 48) from four sub-scores which assess speech and swallowing, (bulbar function), use of upper extremities (cervical function), gait and turning in bed (lumbar function), and breathing (respiratory function). A clinical response is defined as a rate of change of ALSFRS-R of +6 points over 6 months (mean of +1 point per month), where typically patients with ALS have a decline in ALSFRS-R by an average of -1/month.
Time Frame: Pre-Treatment Period (3 months prior to the start of treatment, 2 months prior to the start of treatment, and 1 month prior to the start of treatment), Treatment Period (Day 1 and then monthly until Month 6)
Population: All study participants who received treatment are included in the analysis for this outcome measure, including participants who discontinued treatment early (available ALSFRS-R scores were used).
Measure: Count of Participants; unit: Participants
Groups:
- Immunosuppression Regimen: Participants were monitored for a three month lead-in period prior to beginning treatment. The Baseline Visit 1 occurred within 21 days after the Screening visit and 3 months prior to receiving the first does of the immunosuppressant regimen. Baseline Visits 2 and 3 occurred 2 and 1 month prior to the start of treatment.
  All participants received the same treatment intervention consisting of basiliximab, methylprednisolone, prednisone, tacrolimus and mycophenolate mofetil. Doses of each medication varied by the day of treatment and the treatment period lasted for six months.
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
Participants | 0

2. Secondary Outcome: Mean Rate of Change of ALSFRS-R Scores During Treatment Compared to Pre-Treatment
Description: The ALS Functional Rating Scale - Revised (ALSFRS-R) is an ordinal rating scale (0 through 4) used to determine the ALS patient's self assessment of their ability and need for assistance in 12 activities or functions. This is a validated scale, both in person and by phone, which provides a total score from four sub-scores which assess speech and swallowing, (bulbar function), use of upper extremities (cervical function), gait and turning in bed (lumbar function), and breathing (respiratory function). Total scores range from 0 (most impaired) to 48 (normal ability). ALSFRS-R was measured during the 3 month lead in period and the 6 month treatment period. A random slopes model was fit to the lead-in and treatment periods, with a change point when treatment started. The analysis was based on the difference in slope after the change point. A negative value means that scores during treatment were lower than pre-treatment scores, indicating a decline in ability over time.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale change per month
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
units on a scale change per month | -0.24 (0.23)

3. Secondary Outcome: Mean Rate of Change of Slow Vital Capacity (SVC) During Treatment Compared to Pre-Treatment
Description: Vital capacity (VC), percent of predicted normal, was determined using the slow VC method. SVC measures the amount of air exhaled following a deep breath. For this test, participants hold a mouthpiece in their mouth, breathe in deeply, and breathe out as much air as they can. The test was done seated in a chair and then repeated while lying on an exam table at the Screening Visit. For all other visits, this test was done while seated in a chair. This test takes 15-20 minutes. SVC was measured during the 3 month lead in period and the 6 month treatment period. A random slopes model was fit to the lead-in and treatment periods, with a change point when treatment started. The analysis was based on the difference in slope after the change point. SVC is a way to measure respiratory insufficiency in persons with ALS and SVC decreases as ALS progresses. A negative value means that scores during treatment were lower than pre-treatment scores, indicating a decline over time.
Time Frame: as for outcome 1
Population: All study participants who received treatment are included in the analysis for this outcome measure.
Measure: Mean (Standard Error); unit: percent predicted change per month
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
percent predicted change per month | -0.18 (0.63)

4. Secondary Outcome: Mean Rate of Change of Hand-Held Dynamometry (HHD) During Treatment Compared to Pre-Treatment
Description: Hand held dynamometry (HHD) is a measure of muscle strength and scores decrease as ALS progresses. Six proximal muscle groups were examined bilaterally in both upper and lower extremities. Mean and standard deviation for each muscle group are established from the initial values for each participant. Strength determinations were converted to Z scores and averaged to provide an HHD megascore. The Z-score indicates the number of standard deviations away from the mean of 0. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. HHD was measured during the 3 month lead in period and the 6 month treatment period. A random slopes model was fit to the lead-in and treatment periods, with a change point when treatment started. The analysis was based on the difference in slope after the change point. A negative value means that scores during treatment were lower than pre-treatment scores, indicating a decline in strength over time.
Time Frame: as for outcome 1
Population: All study participants who received treatment are included in the analysis for this outcome measure, including participants who discontinued treatment early.
Measure: Mean (Standard Error); unit: z-score change per month
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
z-score change per month | -0.05 (0.03)

5. Secondary Outcome: Mean Rate of Change in Grip Strength Treatment Compared to Pre-Treatment
Description: Hand grip was measured using a study approved dynamometer to test the maximum isometric strength of the hand and forearm muscles. The grip strength of the left and right hands were analyzed together. Grip strength was measured during the 3 month lead in period and the 6 month treatment period. A random slopes model was fit to the the lead-in and treatment periods, with a change point when treatment started. The analysis was based on the difference in slope after the change point. Grip strength is a measurement of muscle strength and declines as ALS progresses. A positive value means that scores during treatment were higher than pre-treatment scores, indicating an increase in grip strength over time.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: pounds change per month
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
pounds change per month | 1.38 (0.65)

6. Secondary Outcome: Mean Rate of Change of T-cell Subsets in Blood Treatment Compared to Pre-Treatment
Description: Blood was collected for ribonucleic acid (RNA) and the mean rate of decline of T-cells during the 6 month treatment period compared to the pre-treatment period was assessed (blood was collected twice during the 3-month long lead in period). The precise role that T-cells have in ALS is unknown and this study aims to further the understanding of how T-cells operate in persons with ALS. T-cell measurement is a ratio where the relative expression levels of FOXP3 messenger ribonucleic acid (mRNA) was calculated using the Comparative CT Method (ΔΔCT Method), normalizing to β-actin. Samples were obtained during the 3 month lead in period and the 6 month treatment period. A random slopes model was fit to the lead-in and treatment periods, with a change point when treatment started. The analysis was based on the difference in slope after the change point. A negative value means that scores during treatment were lower than pre-treatment scores, indicating a decline in T-cells over time.
Time Frame: Pre-Treatment Period (2 months prior to the start of treatment), Treatment Period (Day 1 and Months 1, 2, 4, 6)
Measure: Mean (Standard Error); unit: fold change per month
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
fold change per month | -0.04 (0.03)

7. Secondary Outcome: Collection of Cerebrospinal Fluid for Future Analysis of Cytokine Levels
Description: Lumbar punctures (LPs) were performed to collect cerebrospinal fluid (CSF). CSF is banked for future use to characterize immune system markers and to further the understanding of the immune factors that contribute to disease progression in ALS. Cytokines are markers of neuroinflammation and can be categorized as neurotoxic or neuroprotective. The role that cytokines play in in ALS progression is still not yet fully understood.
Time Frame: Pre-Treatment Period (two months prior to the start of treatment), Treatment Period (Months 2 and 6), Post-Treatment Period (Month 12)
Population: Cerebrospinal fluid was collected from 29 participants and banked for future analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
Participants | 29

8. Secondary Outcome: Collection of Blood for Future Analysis of Peripheral Blood Mononuclear Cells (PBMCs)
Description: Blood was drawn and banked for future use in order to characterize immune system markers and further the understanding of the immune factors that contribute to disease progression in ALS.
Time Frame: Pre-Treatment Period (2 months prior to the start of treatment), Treatment Period (Day 1 and Months 1, 2, 4, 6), Post-Treatment Period (Months 8 and 12)
Population: Blood was collected for all 31 participants and banked for future use.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppression Regimen
Number analyzed (Participants) | 31
Participants | 31

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events (AEs) from the time they signed the consent form until completion of their participation in the study (defined as death, withdrawal of consent, loss to follow up, early termination due to other reasons, or completion of the entire study).
Description: For the purposes of this study, an adverse event is considered any unfavorable and unintended sign (including clinically significant abnormal laboratory findings), symptom, or disease temporally associated with a study, whether or not the adverse event is considered to be related to the drug product under examination.
Arm/Group | Immunosuppression Regimen
All-Cause Mortality (participants affected / at risk) | 2/31
Serious Adverse Events (participants affected / at risk) | 5/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunosuppression Regimen (N=31)
Hospital admission for dehyration due to dysphagia from ALS (Nervous system disorders) | 1 (1)
Hospitalization due to knee injury from a fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Hospitalization due to a kidney stone (Renal and urinary disorders) | 1 (1)
Hospitalization due to pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization due to bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Asymptomatic T-wave inversions with troponin elevation (Cardiac disorders) | 1 (1) — Asymptomatic T-wave inversions with slight troponin elevation; no indication of an acute cardiac event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunosuppression Regimen (N=31)
Fall (General disorders) | 17 (48)
Diarrhea (Gastrointestinal disorders) | 13 (17)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 12 (27)
Headache (General disorders) | 11 (16)
Muscular Spasms (Musculoskeletal and connective tissue disorders) | 11 (14)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Nausea (General disorders) | 4 (5)
Cold Sore (Infections and infestations) | 1 (4)
Tracheal bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal insufficiency (elevated creatinine) (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes